CLINICAL TRIAL: NCT01263756
Title: A Study of the Driving Performance of Individuals With Autism Spectrum Disorders
Brief Title: Autism Spectrum Disorders (ASD) Driving Study
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief of the Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Other Study IDs: 2010-P-000173
Record Dates: First submitted 2010-11-29; First posted 2010-12-21 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Driving; Autism Spectrum Disorders; ASD; Attention Deficits; Adults; Adolescents; Pervasive Developmental Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ASD group: Adolescents and adults with Autism Spectrum Disorders (ASDs).

SUMMARY:
The proposed pilot study will begin to assess whether driving impairments are included in the functional deficits associated with Autism Spectrum Disorders (ASDs). This will be completed by obtaining data on velocity, collision risk, and visual attention of subjects with ASDs who drive in a simulator. The study includes 2-3 visits for the screening period (approximately 6 hours of assessments) and one driving simulation visit (approximately 2.5 hours). The investigators expect to enroll 20 adolescents and adults (ages 16-50, inclusive) who have been identified as having an ASD from a prior diagnosis or participation in community conferences for individuals with ASDs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 16-50 years
* Identification as having ASD from a prior diagnosis or participation in community conferences for individuals with ASD

Exclusion Criteria:

* Major sensorimotor handicaps (e.g. deafness, blindness)
* Inadequate command of the English language
* Individuals who have never held a valid driver's license
* Mental retardation (IQ < 80)

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and adults, ages 16-50, with Autism Spectrum Disorders.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Simulated driving performance of adolescents and adults with ASDs. | one-time observation (3 hour assessment)
  Data will be obtained on velocity, collision risk, and visual attention of subjects with ASDs who drive in the driving simulator at the Massachusetts Institute of Technology (MIT).

SECONDARY OUTCOMES:
Questionnaire measures of driving history and behavior of adolescents and adults with ASDs. | one-time assessment (2-6 hour screening visit)
  Subjects with ASD will complete two questionnaires, the Driver Behavior Questionnaire and the Driving History Questionnaire, to provide data on the frequency of violations, errors, accidents, and other aspects of driving history and behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States